CLINICAL TRIAL: NCT05240781
Title: Zotarolimus Eluting Stent Versus Sirolimus Eluting Stent in High Bleeding Risk Angioplasty
Brief Title: Zotarolimus vs Sirolimus Eluting Stent in High Bleeding Risk
Acronym: ZEVS-HBR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Daniel Fernando Zazueta Salido, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-1277
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: High Bleeding Risk; Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Short DAPT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, non-inferiority clinical trial enrolling eligible subjects with high bleeding risk and coronary artery disease to be treated by percutaneous coronary intervention at the National Institute of Cardiology "Ignacio Chávez" in México. Included patients will have follow-up at the outpatient clinic through 1 year, until death or study exit, whichever comes first.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized treatment will not be revealed to patient or data analyst at any time during procedure or afterwards until follow-up and analysis has been done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zotarolimus Eluting Stent (Active Comparator): High Bleeding Risk patients to be treated with drug-eluting stents (DES). Includes both stable Coronary Artery Disease (CAD) and Acute Coronary Syndrome (ACS) patients undergoing elective PCI.
  Interventions: Device: Zotarolimus eluting stent
- Sirolimus Eluting Stent (Experimental): High Bleeding Risk patients to be treated with drug-eluting stents (DES). Includes both stable CAD and ACS patients undergoing elective PCI.
  Interventions: Device: Sirolimus eluting stent

INTERVENTIONS:
Device: Zotarolimus eluting stent — Size (diameter and length) will be chosen at operator's discretion aided by simple angiography, QCA, or intravascular image; so that the lesion previously prepared and 2 mm at each end are covered by DES with an stent to artery ratio of 1.1. Post-dilatation will be performed when indicated. Device will be used by CE mark instructions.
  All patients will receive DAPT as follows: After a loading dose (if necessary) of aspirin and a P2Y12 inhibitor, aspirin 100 mg and a P2Y12 inhibitor daily will be indicated for 1 month in both ACS and Chronic Coronary Syndrome (CCS). Patients with high ischemic risk could be extended to 3 months. After DAPT, SAPT will be continued with the drug of choice, preferably P2Y12 inhibitor. Patients requiring chronic anticoagulation will receive triple therapy only during hospitalization. At release, an oral anticoagulant (NOAC preferred over VKA) will be indicated along with 6 months of SAPT with a P2Y12 inhibitor.
  Other Names: Resolute Onyx, Zotarolimus eluting stent (Medtronic, Santa Rosa, CA, USA)
  Arms: Zotarolimus Eluting Stent
Device: Sirolimus eluting stent — Size (diameter and length) will be chosen at operator's discretion aided by simple angiography, QCA, or intravascular image; so that the lesion previously prepared and 2 mm at each end are covered by DES with an stent to artery ratio of 1.1. Post-dilatation will be performed when indicated. Device will be used in accordance with the CE mark instructions.
  All patients will receive DAPT as follows: After a loading dose (if necessary) of aspirin and a P2Y12 inhibitor, aspirin 100 mg and a P2Y12 inhibitor daily will be indicated for 1 month in both ACS and CCS. Patients with high ischemic risk could be extended to 3 months. After DAPT, SAPT will be continued with the drug of choice, preferably P2Y12 inhibitor. Patients requiring chronic anticoagulation will receive triple therapy only during hospitalization. At release, an oral anticoagulant (NOAC preferred over VKA) will be indicated along with 6 months of SAPT with a P2Y12 inhibitor.
  Other Names: Ultimaster, Sirolimus eluting stent (Terumo; Tokyo, Japan); Ultimaster Tansei, Sirolimus eluting stent (Terumo; Tokyo, Japan)
  Arms: Sirolimus Eluting Stent

SUMMARY:
Randomized, single-blind, single-center, non-inferiority clinical trial to compare target lesion failure (TLF) at 12 months in high bleeding risk patients who underwent elective coronary percutaneous intervention with a zotarolimus eluting stent versus a sirolimus eluting stent and short Dual Antiplatelet Therapy (DAPT).

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years old or older with an ischemic de-novo lesion(s) in coronary artery or coronary bypass graft suitable for percutaneous coronary intervention, in context of acute coronary syndrome or chronic coronary syndrome with evidence of ischemia by non-invasive study or pressure guidewire that can be treated by DES, and has at least 1 major or 2 minor Academic Research Consortium High Bleeding Risk criteria:

Major criteria:

* 1. Anticipated use of long-term oral anticoagulation
* 2. Severe or end-stage Chronic Kidney Disease (CKD) (eGFR <30 mL/min)
* 3. Hemoglobin < 11 g/dL
* 4. Spontaneous bleeding requiring hospitalization or transfusion in the last 6 months, or any time, if recurrent.
* 5. Moderate or severe baseline thrombocytopenia (<100,000/uL)
* 6. Chronic bleeding diathesis
* 7. Liver cirrhosis with portal hypertension
* 8. Active malignancy (excluding nonmelanoma skin cancer) within the past 12 months
* 9. Previous spontaneous intracranial hemorrhage
* 10. Previous traumatic intracranial hemorrhage within the past 12 months
* 11. Presence of Brain Arteriovenous malformation (AVM)
* 12. Moderate or severe ischemic stroke (NIHSS score equal or more than 5) within the past 6 months
* 13. Non-deferrable major surgery on DAPT
* 14. Recent major surgery or major trauma within 30 days before PCI

Minor Criteria:

* 1. Age 75 years old and older
* 2. Moderate CKD (eGFR 30-59 mL/min)
* 3. Hemoglobin 11 - 12.9 g/dL in men and 11 - 11.9 g/dL in women
* 4. Spontaneous bleeding requiring hospitalization or transfusion within the past 12 months, not meeting major criterion
* 5. Long term use of NSAIDs or steroids
* 6. Any ischemic stroke at any time not meeting major criterion

Exclusion Criteria:

* STEMI undergoing primary PCI
* Cardiogenic shock or resuscitation with uncertain neurological status at arrival to PCI
* Unprotected left main lesion
* Reference diameter larger or shorter than available stents
* Life expectancy < 12 months
* In-stent restenosis o thrombosis of previous stent
* Inability to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Rate of composed of cardiovascular death, myocardial infarction related to the treated vessel or ischemia driven target lesion revascularization

SECONDARY OUTCOMES:
Cardiovascular death | 12 months
  Rate of death resulting from cardiovascular causes:
  Death caused by acute MI Death caused by sudden cardiac, including unwitnessed, death Death resulting from heart failure Death caused by stroke Death caused by cardiovascular procedures Death resulting from cardiovascular hemorrhage Death resulting from other cardiovascular cause Any MI not clearly attributable to a non- target vessel will be considered as target-vessel MI.
  Percutaneous coronary intervention (PCI) related MI is termed type 4a MI.
Myocardial Infarction related to the treated vessel | 12 months
  Rate of myocardial infarction related to the treated vessel (according to the 4th international definition of myocardial infarction): detection of an increase or decrease in cardiac troponin values with at least 1 of the values above the upper reference limit of the 99th percentile and at least 1 of the following conditions :
  Symptoms of acute myocardial ischemia. New ischemic changes in the electrocardiogram. Appearance of pathological Q waves. Imaging evidence of loss of viable myocardium or new regional abnormalities in myocardial wall mobility following a pattern compatible with ischemic etiology.
  Identification of a coronary thrombus by angiography with intracoronary imaging or by autopsy Any MI that cannot be clearly attributed to a vessel other than the revascularized one will be considered as MI related to the treated vessel.
Target Lesion Revascularization | 12 months
  Rate of repeated percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Target Vessel Failure (TVF) | 12 months
  Rate of TVF (composed of cardiovascular death, myocardial infarction related to the treated vessel or ischemia driven target vessel revascularization)
Target Vessel Revascularization | 12 months
  Rate of repeat percutaneous intervention or surgical bypass of any segment of the target vessel
Non-cardiovascular death | 12 months
  Rate of any death that is not thought to be the result of a cardiovascular cause:
  1. Death resulting from malignancy
  2. Death resulting from pulmonary causes
  3. Death caused by infection (includes sepsis)
  4. Death resulting from gastrointestinal causes
  5. Death resulting from accident/trauma
  6. Death caused by other noncardiovascular organ failure 7. Death resulting from other noncardiovascular cause
Major Bleeding | 12 months
  Incidence of bleeding complications according to The Bleeding Academic Research Consortium 2 (BARC-2) scale: 3 or greater
Technical success | Periprocedural
  Rate of restoration of antegrade Thrombolysis In Myocardial Infarction (TIMI) flow 2 or 3 and a <30% residual stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Guering Eid-Lidt, MD, Study Director — Instituto Nacional de Cardiología "Ignacio Chávez"; Daniel F Zazueta, MD, Principal Investigator — Instituto Nacional de Cardiología "Ignacio Chavez"
Locations (1):
- Instituto Nacional de Cardiología "Ignacio Chávez", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa F, Van Klaveren D, Feres F, James S, Raber L, Pilgrim T, Hong MK, Kim HS, Colombo A, Steg PG, Bhatt DL, Stone GW, Windecker S, Steyerberg EW, Valgimigli M; PRECISE-DAPT Study Investigators. Dual Antiplatelet Therapy Duration Based on Ischemic and Bleeding Risks After Coronary Stenting. J Am Coll Cardiol. 2019 Feb 26;73(7):741-754. doi: 10.1016/j.jacc.2018.11.048. PMID 30784667
- [Background] Costa F, Tijssen JG, Ariotti S, Giatti S, Moscarella E, Guastaroba P, De Palma R, Ando G, Oreto G, Zijlstra F, Valgimigli M. Incremental Value of the CRUSADE, ACUITY, and HAS-BLED Risk Scores for the Prediction of Hemorrhagic Events After Coronary Stent Implantation in Patients Undergoing Long or Short Duration of Dual Antiplatelet Therapy. J Am Heart Assoc. 2015 Dec 7;4(12):e002524. doi: 10.1161/JAHA.115.002524. PMID 26643501
- [Background] Urban P, Mehran R, Colleran R, Angiolillo DJ, Byrne RA, Capodanno D, Cuisset T, Cutlip D, Eerdmans P, Eikelboom J, Farb A, Gibson CM, Gregson J, Haude M, James SK, Kim HS, Kimura T, Konishi A, Laschinger J, Leon MB, Magee PFA, Mitsutake Y, Mylotte D, Pocock S, Price MJ, Rao SV, Spitzer E, Stockbridge N, Valgimigli M, Varenne O, Windhoevel U, Yeh RW, Krucoff MW, Morice MC. Defining High Bleeding Risk in Patients Undergoing Percutaneous Coronary Intervention. Circulation. 2019 Jul 16;140(3):240-261. doi: 10.1161/CIRCULATIONAHA.119.040167. Epub 2019 May 22. PMID 31116032
- [Background] Varenne O, Cook S, Sideris G, Kedev S, Cuisset T, Carrie D, Hovasse T, Garot P, El Mahmoud R, Spaulding C, Helft G, Diaz Fernandez JF, Brugaletta S, Pinar-Bermudez E, Mauri Ferre J, Commeau P, Teiger E, Bogaerts K, Sabate M, Morice MC, Sinnaeve PR; SENIOR investigators. Drug-eluting stents in elderly patients with coronary artery disease (SENIOR): a randomised single-blind trial. Lancet. 2018 Jan 6;391(10115):41-50. doi: 10.1016/S0140-6736(17)32713-7. Epub 2017 Nov 1. PMID 29102362
- [Background] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Background] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Palmerini T, Bacchi Reggiani L, Della Riva D, Romanello M, Feres F, Abizaid A, Gilard M, Morice MC, Valgimigli M, Hong MK, Kim BK, Jang Y, Kim HS, Park KW, Colombo A, Chieffo A, Ahn JM, Park SJ, Schupke S, Kastrati A, Montalescot G, Steg PG, Diallo A, Vicaut E, Helft G, Biondi-Zoccai G, Xu B, Han Y, Genereux P, Bhatt DL, Stone GW. Bleeding-Related Deaths in Relation to the Duration of Dual-Antiplatelet Therapy After Coronary Stenting. J Am Coll Cardiol. 2017 Apr 25;69(16):2011-2022. doi: 10.1016/j.jacc.2017.02.029. PMID 28427576
- [Background] Xu XM, Vestesson E, Paley L, Desikan A, Wonderling D, Hoffman A, Wolfe CD, Rudd AG, Bray BD. The economic burden of stroke care in England, Wales and Northern Ireland: Using a national stroke register to estimate and report patient-level health economic outcomes in stroke. Eur Stroke J. 2018 Mar;3(1):82-91. doi: 10.1177/2396987317746516. Epub 2017 Nov 30. PMID 29900412
- [Result] Windecker S, Latib A, Kedhi E, Kirtane AJ, Kandzari DE, Mehran R, Price MJ, Abizaid A, Simon DI, Worthley SG, Zaman A, Hudec M, Poliacikova P, Abdul Ghapar AKB, Selvaraj K, Petrov I, Mylotte D, Pinar E, Moreno R, Fabbiocchi F, Pasupati S, Kim HS, Aminian A, Tie C, Wlodarczak A, Hur SH, Marx SO, Jankovic I, Brar S, Bousquette L, Liu M, Stone GW; ONYX ONE Investigators. Polymer-based or Polymer-free Stents in Patients at High Bleeding Risk. N Engl J Med. 2020 Mar 26;382(13):1208-1218. doi: 10.1056/NEJMoa1910021. Epub 2020 Feb 12. PMID 32050061
- [Result] Valgimigli M, Frigoli E, Heg D, Tijssen J, Juni P, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Tonino PAL, Roffi M, Lesiak M, Mahfoud F, Bartunek J, Hildick-Smith D, Colombo A, Stankovic G, Iniguez A, Schultz C, Kornowski R, Ong PJL, Alasnag M, Rodriguez AE, Moschovitis A, Laanmets P, Donahue M, Leonardi S, Smits PC; MASTER DAPT Investigators. Dual Antiplatelet Therapy after PCI in Patients at High Bleeding Risk. N Engl J Med. 2021 Oct 28;385(18):1643-1655. doi: 10.1056/NEJMoa2108749. Epub 2021 Aug 28. PMID 34449185